CLINICAL TRIAL: NCT06961370
Title: A Phase I, Multi-center, Multi-part Study to Investigate Safety, Tolerability, PK, PD, and Immunogenicity of RO7669330 Intravitreal Injections in Participants With GA Secondary to AMD: Part 1A: Open-label, MAD; Part 1B: Randomized PD Pilot; Part 2: Masked, Randomized, Active-comparator-controlled
Brief Title: A Study to Investigate Safety, Tolerability, Pharmacokinetics (PK), Pharmacodynamics (PD), and Immunogenicity of RO7669330 in Participants With Geographic Atrophy (GA) Secondary to Age-related Macular Degeneration (AMD)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BP45482
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Geographic Atrophy; Age-related Macular Degeneration
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration | interventions — pegcetacoplan

STUDY DESIGN:
Intervention Model Description: Part 1A will be a single group study, while Part 1B and Part 2 will follow a parallel-group design.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Part 1A of the study will be open-label and non-randomized while Part 1B and 2 will be masked and randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1A: Multiple Ascending Dose (MAD) (Experimental): Participants will receive multiple doses of RO7669330 as IVT injections in the study eye with additional cohorts of participants receiving higher doses of RO7669330.
  Interventions: Drug: RO7669330
- Part 1B: Syfovre and Izervay (Experimental): Participants will receive either Syfovre, 15 milligrams (mg) or Izervay, 2 mg, as an IVT injection in the study eye.
  Interventions: Drug: Syfovre™; Drug: Izervay™
- Part 2: RO7669330 vs Active Comparator (Syfovre or Izervay) (Experimental): Participants will receive RO7669330 (at two dose levels) or the active comparator (either Syfovre or Izervay), as an IVT injection in the study eye.
  Interventions: Drug: RO7669330; Drug: Syfovre™; Drug: Izervay™

INTERVENTIONS:
Drug: RO7669330 — RO7669330 will be administered as an IVT injection in the study eye per the schedule specified in the respective arms.
  Arms: Part 1A: Multiple Ascending Dose (MAD); Part 2: RO7669330 vs Active Comparator (Syfovre or Izervay)
Drug: Syfovre™ — Syfovre™ will be administered as an IVT injection in the study eye per the schedule specified in the respective arms.
  Other Names: Pegcetacoplan injection
  Arms: Part 1B: Syfovre and Izervay; Part 2: RO7669330 vs Active Comparator (Syfovre or Izervay)
Drug: Izervay™ — Izervay™ will be administered as an IVT injection in the study eye per the schedule specified in the respective arms.
  Other Names: Avacincaptad pegol IVT solution
  Arms: Part 1B: Syfovre and Izervay; Part 2: RO7669330 vs Active Comparator (Syfovre or Izervay)

SUMMARY:
The main purpose of this study is to assess the ocular and systemic safety and tolerability of RO7669330 in participants with GA secondary to AMD in at least one eye in Part 1, or both eyes in Part 2, after multiple unilateral intravitreal (IVT) doses.

ELIGIBILITY:
Inclusion Criteria:

* Adequately clear ocular media, adequate pupillary dilation, and fixation to allow acquisition of good quality fundus imaging
* GA that resides completely within the fundus autofluorescence (FAF) imaging field
* Presence of hyperautofluorescence of either banded or diffuse pattern adjacent to the GA area on FAF
* Study eye has early treatment of diabetic retinopathy study (ETDRS) best-corrected visual acuity (BCVA) score as follows:
* Part 1A: 19 to 48 letters, inclusively
* Part 1B: > 19 letters
* Part 2: ≥ 24 letters
* Total GA lesion size must be as follows:
* Parts 1A and 1B: ≥ 1.25 square millimeter (mm^2) and ≤ 20 mm^2 )
* Part 2: ≥ 2.5 mm^2 and ≤ 20 mm^2

Exclusion Criteria:

Ocular Exclusion Criteria for the Study Eye:

* Aphakic or pseudophakic with intraocular lens outside of the capsular bag
* Previous laser photocoagulation or IVT anti-vascular endothelial growth factor (VEGF) for CNV, diabetic macular edema (DME), retinal vein occlusion (RVO), or proliferative diabetic retinopathy
* Active or history of CNV

Ocular Exclusion Criteria for the Non-Study Eye:

- Non-functioning non-study eye, defined as either: BCVA of hand motion or worse and/or no physical presence of eye

Ocular Exclusion Criteria for Both Eyes:

* Macular atrophy in either eye due to causes other than AMD
* Part 2: Evidence of prior or active CNV
* Prior treatment with any approved therapy for GA (Syfovre, Izervay) in either eye for Part 1A and Part 2 ≤ 20 weeks prior to Day 1. For Part 1B, prior treatment with any approved therapy for GA (Syfovre, Izervay) in the study eye ≤ 20 weeks prior to Day 1

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2027-01-03 (Estimated); Study Completion 2027-01-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Up to a maximum of 34 weeks
Number of Participants With Abnormalities Recorded in Standard Ophthalmological Assessments | Up to a maximum of 34 weeks
  The standard ophthalmological assessments that will be conducted may include the following: slit-lamp, indirect ophthalmology, intraocular pressure (IOP), best corrected visual acuity (BCVA), spectral domain optical coherence tomography (SD-OCT), fundus fluorescein angiography (FFA), and color fundus photography (CFP).

SECONDARY OUTCOMES:
Part 1A and Part 2: Ocular and Systemic Concentration of RO7669330 | Up to a maximum of Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (16):
- United States (16):
  - Associated Retina Consultants - Phoenix - DocTrials - PPDS, Phoenix, Arizona
  - Barnet Dulaney Perkins Eye Center, Sun City, Arizona
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Global Research Management, Glendale, California
  - Retinal Consultants Medical Group Inc - Parkcenter Drive, Sacramento, California
  - Southeast Retina Center, Augusta, Georgia
  - Cumberland Valley Retina Consultants PC, Hagerstown, Maryland
  - The Retina Institute, St Louis, Missouri
  - Retina Northwest, Portland, Oregon
  - Erie Retina Research, Erie, Pennsylvania
  - Charles Retina Institute, Germantown, Tennessee
  - Tennessee Retina PC, Nashville, Tennessee
  - Austin Clinical Research, LLC, Austin, Texas
  - Texas Retina Associates, Dallas, Texas
  - Retina Consultants of Texas Westover Hills Retina Center, San Antonio, Texas
  - Retina Consultants of Texas - (The Woodlands), The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No